CLINICAL TRIAL: NCT07024628
Title: Heat Smart: Empowering Primary Care Providers to Safeguard Vulnerable Populations Against Extreme Heat
Brief Title: Assessing the Effectiveness of Heat Adaptation Digital Messages From Primary Care Providers to Their Patients on the Change in Behaviour for Heatwave-related Preparedness
Acronym: HeatSmart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Montfort (Other)
Collaborators: Children's Hospital of Eastern Ontario Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 24-25-02-055
Record Dates: First submitted 2025-05-28; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Heathly Subjects; Primary Health Care; Climate Change; Public Health; Preventive Health Services (PREV HEALTH SERV); Environmental Exposure; Risk Reduction Behavior; Heat Stress Disorders; Heat Exposure
Keywords: primary care; digital messaging; heatwave; climate change; public health; CPIN
MeSH Terms: conditions — Risk Reduction Behavior; Heat Stress Disorders

STUDY DESIGN:
Intervention Model Description: This study employs a cluster randomized controlled trial (RCT) to evaluate the impact of a heat adaptation digital messages intervention. Only primary care practices with at least 2 participating practitioners will be included in the study, where each PCP will act as a patient cluster. For each practice, the Primary Care Providers will be randomly assigned, and all their adult patient panel will either receive heat smart adaptation digital messages (the exposed group) or non-heat wave health promotion digital messages (the control group).
  There will be continuous recruitment through the study. Outcomes will be assessed after each heatwave. This means that participants enrolled at the start of the study will have a greater number of timepoints for data collection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated - receive heat adaptation digital messages (Experimental): Patients in the Treated arm will receive messages to equip and prepare them for extreme heat events. The intervention is multifaceted: the first message will to encourage patients to prepare by creating a heat safety plan, and to form Check-in Companion groups among friends, neighbours, and relatives as well as to connect patients with existing key infrastructure that can be vital during heat events (ex: cooling stations and public facilities with air conditioning).
  When a heat-advisory is announced, additional messages will be sent to alert patients in the Treated group to activate their heat safety plans.
  Interventions: Other: Heat adaptation digital messaging
- Control (Active Comparator): Patients in the Control arm will receive messages not related to heat waves. These messages will be related to other environmental risks
  Interventions: Other: Non-heat-related digital messaging

INTERVENTIONS:
Other: Heat adaptation digital messaging — Digital messages to equip and prepare patients for extreme heat events. The first message will to encourage patients to prepare by creating a heat safety plan, and to form Check-in Companion groups among friends, neighbours, and relatives as well as to connect patients with existing key infrastructure that can be vital during heat events (ex: cooling stations and public facilities with air conditioning). When a heat-advisory is announced, additional messages will be sent to alert patients in the Treated group to activate their heat safety plans.
  Arms: Treated - receive heat adaptation digital messages
Other: Non-heat-related digital messaging — Digital health promotion messages not related to heatwaves
  Arms: Control

SUMMARY:
Extreme heat events pose a significant health threat in Canada, as demonstrated by the 2021 heat wave that claimed over 600 lives in Western Canada. Most heat-related deaths occur indoors and are preventable. Primary care providers (PCPs), who serve 88% of Canadians, are uniquely positioned to identify and support at-risk individuals. Heat Smart, in alignment with Heat Alert and Response Systems (HARS), aims to bridge the gap between primary care and public health to enhance community resilience and reduce health inequities related to extreme heat events.

This randomized control trial in Eastern Ontario will examine whether patients receiving tailored digital health messages from their family physician or nurse practitioner change their behaviour to protect themselves from extreme heat-related illness. The Heat Smart study will:

* Assess risk: Analyze electronic medical records and patient surveys to identify vulnerable individuals.
* Deliver tailored messages: Send personalized digital guidance via e-mail or text, offering heat safety advice and local resource information in English and French.
* Issue early warning alerts: Notify at-risk patients of upcoming heat events, prompting action.
* Evaluate impact: Use surveys and health data to measure effectiveness in reducing heat-related health impacts.

Short-term outcomes include increased awareness and preparedness among patients about heat-related health risks. Long-term goals involve scaling the intervention across Canada to reduce heat-related illnesses, enhance social connectedness, and decrease healthcare utilization.

DETAILED DESCRIPTION:
Primary Hypothesis

The study will test the following primary hypothesis: "Patients who receive tailored digital health promotion messages from their primary care providers will perform more heat adaptive proactive behaviours to protect themselves from heat-related illness compared to those who do not receive such messages."

Secondary Hypotheses

1. Patients receiving Heat Smart messages will demonstrate greater engagement in specific heat preparedness activities, such as creating heat safety plans and forming networks among friends, neighbours, and relatives (patient survey data).
2. Patients in the intervention group will experience lower rates of heat-related healthcare utilization, as measured by primary care provider visits, emergency department visits and filling prescription drugs during heat events (ICES data).
3. The intervention will be effective across different socio-demographic subpopulations, including older adults, individuals with chronic illnesses, and socially isolated individuals.
4. The integration of primary care into HARS will enhance public health system coordination and improve response strategies for extreme heat events.

This study employs a cluster randomized controlled trial (RCT) to evaluate the impact of a heat adaptation digital messages intervention. Only primary care practices with at least 2 participating practitioners will be included in the study, where each PCP will act as a patient cluster. For each practice, the Primary Care Providers will be randomly assigned, and all their adult patient panel will either receive heat smart adaptation digital messages (the exposed group) or non-heat wave health promotion digital messages (the control group).

The study follows an intention-to-treat (ITT) design, meaning that all participants who consent to participate will be analyzed based on their original group assignment, regardless of adherence to the heat smart digital messages intervention (e.g., did the participant read the message). The study will have a two-year follow-up period to assess behavioural changes related to heat adaptation.

Research Objectives

The Heat Smart project aims to enhance primary care involvement in public health led heat adaptation strategies and improve the preparedness of at-risk populations for extreme heat events.

1. Assess Individual-Level Risks for Excessive Heat-Related Illnesses

   * Identify patients at increased risk of heat-related illness using primary care provider's electronic medical records and patient surveys.
   * Characterize socio-cultural, demographic, and clinical factors that contribute to heat vulnerability, including:

     * Age (older adults, children)
     * Chronic illnesses (e.g., cardiovascular disease, diabetes, asthma, mental health conditions)
     * Social isolation and poverty
     * Use of medications that impair thermoregulation
   * Segment patients into subpopulations based on shared characteristics to tailor interventions.
   * Assess patients' information needs and barriers to heat preparedness.
2. Implement and Evaluate a Digital Messaging Intervention

   * Deliver tailored, evidence-based digital messages (via email or text) to all adult patients of participating primary care providers to:

     * Educate them on heat-related health risks.
     * Encourage the development of personalized heat safety plans for patients at increased risk.
     * Provide information about local cooling stations, transportation options, and emergency resources.
   * Issue early warning alerts to at-risk patients when excessive heat events are imminent.
   * Evaluate the impact of the intervention through:

     * Patient surveys assessing self-reported behaviour change in heat preparedness.
     * Linking patient survey responses to health administrative data to measure healthcare utilization (e.g., emergency department visits, prescription medication use).
   * Determine the effectiveness of integrating primary care providers into public health-led Heat Alert and Response Systems (HARS).
3. Scale and Expand the Intervention

   * Refine and adapt the intervention based on rapid-cycle evaluations.
   * Expand to two additional provinces to test scaling feasibility.
   * Develop a national model for integrating primary care into climate adaptation strategies, ensuring scalability and sustainability.
4. Improve Health Equity and Climate Resilience

   * Target vulnerable and equity-deserving populations, ensuring that interventions are tailored to their needs.
   * Encourage social connectedness by fostering Check-in Companion heat response groups among friends, neighbours, and relatives.
   * Enhance collaboration between primary care and public health to create a cohesive, system-wide approach to adaptation to extreme heat events.
   * Provide policy-relevant insights to inform national heat adaptation strategies and reduce health inequities.

These objectives align with Canada's HeatADAPT Program and National Adaptation Strategy, ensuring a whole-of-society approach to protecting health during extreme heat events.

Randomization

* Patients will be assigned to intervention or control arms using cluster randomization. Block of sizes of 2 will be used to randomly assign the primary care provider to either the treatment or control arms, to ensure balance between groups and between practices.
* After randomization, balance across the two arms will be assessed using variables associated with vulnerability (e.g., age, sex, housing marginalization (ONT-Marg, based on 6-digit postal code) is included as a covariate to account for socio-economic disparities in vulnerability to heat-related events, neighbourhood rurality, self-reported baseline Heat Action Plan, chronic illness (e.g., cardiovascular disease, diabetes, asthma, mental health conditions) and heat susceptible diseases (e.g., requiring medications that impair thermoregulation)).

ELIGIBILITY:
Inclusion Criteria:

The Heat Smart randomized controlled trial study will recruit patients and primary care providers (PCPs) from Eastern Ontario. The inclusion criteria ensure that the intervention reaches at-risk individuals while being scalable across different patient populations:

Primary Care Patients:

* Adults (18 years and older)
* Patients must be registered with a participating PCP.
* They must have had at least one visit with their PCP in the past two years to ensure active engagement.
* Participants must have an active email, cell phone or messaging service (SMS) to receive Heat Smart digital messages.
* Patients must be able to understand and consent to participate in the study.
* Patients must be able to communicate in at least one of the official languages (English, French).
* Participants will be recruited from PCP located in two Eastern Ontario public health districts: the Eastern Ontario Health Unit and Ottawa Public Health (including urban, rural, and Indigenous communities such as Akwesasne).

Primary Care Providers:

* Must be a licensed Family Physician (FP) or Nurse Practitioner (NP) in a practice of at least 2 PCPS.
* The providers must be offering comprehensive primary care to a panel of patients (not solely urgent care or walk-in services).
* Must work in a computerized primary care clinic with an electronic medical record system.
* Must expect to remain in practice for at least 24 months.
* Must be located in Eastern Ontario.
* Must be willing to use the Canadian Primary Care Information Network (CPIN) to deliver Heat Smart messages and surveys.
* Must be using Cliniconex or Qualtrics as a practice tool for communication enabling outreach before the patients are invited to consent to participate in the study.

Exclusion Criteria:

Patients who do not read French or English will be excluded from the study as they will not be able to give informed consent or to fill out the surveys. Patients who do not have an email address or text messaging service will be excluded for the same reason. Minors, patients with dementia and people who cannot read and write in English or French will not be eligible because the automated approach to surveying patients makes it impractical to properly obtain their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who report adopting at least one heat adaptation behaviour via self-report survey | Assessed after a heatwave event, up to 2 years following enrollment.
  Participants will be asked: "Have you taken any action to prepare for a heat wave?" (yes/no).

SECONDARY OUTCOMES:
Number of heat-adaptation behaviours self-reported by the participants. | Assessed after a heatwave event, up to 2 years following enrollment.
  Participants will be asked a question about which heat-adaptive behaviours they undertook prior to the most recent heat wave.

OTHER OUTCOMES:
Self-reported heatwave-related challenges: frequency of economic and lifestyle impacts | Assessed after a heatwave event, up to 2 years following enrollment.
  Participants will select from a list of impacts (e.g., missed work, medical costs, utility bills, missed activities, increased caregiving responsibilities). Results will be reported as the proportion selecting each option.
Heatwave health risk and preparedness beliefs - Likert scores | Assessed after a heatwave event, up to 2 years following enrollment.
  Participants will respond to three belief statements on a 5-point Likert scale (1 = Strongly Disagree, 5 = Strongly Agree):
  1. If I do not take steps to cool my home, keep my body cool, or stay hydrated during a heatwave, I may experience a medical emergency
  2. I believe I have the resources and information needed to avoid a medical emergency during a heatwave.
  3. Staying in touch with someone during a heatwave is important for my health.
Frequency of social interactions during heatwaves | Assessed after a heatwave event, up to 2 years following enrollment.
  Participants will report number of in-person or virtual interactions during the most recent heatwave using categorical options (none; 1-3; 4-6; 7+). Responses will be summarized as proportions by category.
Knowledge of heat waves - score based on number of correct answers | Assessed after a heatwave event, up to 2 years following enrollment.
  Four true/false questions assessing understanding of the health risks of heatwaves

CONTACTS AND LOCATIONS:
Locations (1):
- Institut du Savoir Montfort, Ottawa, Ontario, Canada